CLINICAL TRIAL: NCT02027818
Title: Study of the (Intravenously Injected) Indocyanine Green Distribution in the Margins of Breast Cancer After Tumorectomy
Brief Title: Study of the ICG Distribution in the Margins of Breast Cancer After Tumorectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BR-TUM-ICG-IV
Record Dates: First submitted 2014-01-02; First posted 2014-01-06 (Estimated); Last update posted 2023-12-15 (Actual); Status verified 2013-12

CONDITIONS: Breast Cancer
Keywords: margins; tumorectomy
MeSH Terms: conditions — Breast Neoplasms; Margins of Excision | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Indocyanine Green (Experimental): study of the correlation between fluorescence and margins of the tumours after iv injection of Indocyanine Green
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — Observation of the correlation between fluorescence and margins of the tumour after IV injection of ICG
  Other Names: ICG

SUMMARY:
We will observe if ICG fluorescence correlates with margins of breast tumours after iv injection of the contrast agent

DETAILED DESCRIPTION:
In the operating room:

ICG 0.25 mg/kg will be given as an iv injection at least 20 minutes before the beginning of the operation.

The surgeon will remove the tumour (and the axillary lymph nodes) as usual.

Optionally, peroperative "in vivo" imaging of the dissection of the tumour using the PDE camera will be performed.

In the Laboratory of Pathology:

The "fresh" tumorectomy piece will be processed as usual, and the thick sections for the evaluation of the margins as well as the tissues samples from each margins will be imaged using the PDE in comparison with the fluorescence in the mid part of the tumour and the fluorescent areas will be so delimited (and later analyzed in comparison with standards of known fluorescence intensity).

After fixation, the tumoral tissues will be thereafter processed "as usual".

If fluorescent foci are identified at the level of the axillary piece (in case of CALND), they will be dissected and processed as other lymph nodes. Additionally, metastatic lymph nodes -if present- will also be controlled for their microscopic fluorescence or not.

Using the near-infrared fluorescence microscope, the slides corresponding to the macroscopically fluorescent structures will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histopathological diagnosis of mammary cancer who are candidate for tumorectomy, either with SLN selective lymphadenectomy, or with complete axillary node dissection,
* Informed consent form signed.

Exclusion Criteria:

* Diagnosis of mammary cancer established by "gross" biopsy,
* Age less than18 years old.
* Inability to give informed consent.
* History of allergy or hypersensitivity against the investigational product (its active substance or ingredients), to iodine or to shellfish.
* Apparent hyperthyroidism, autonomous thyroid adenoma, unifocal, multifocal or disseminated autonomies of the thyroid gland.
* Documented coronary disease.
* Advanced renal impairment (creatinine > 1,5mg/dl).
* During the 2 weeks before the enrolment, concurrent medication which reduces or increases the extinction of ICG (i.e. anticonvulsants, haloperidol and Heparin).
* Pregnancy, breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
- Evaluation of the ability of NIR imaging to show (fluorescent) the tumoral volumes, the tumoral tissues to be analyzed by the pathologist, especially at the level of the operative margins | 17 months

SECONDARY OUTCOMES:
- Analysis of the correlation between (levels of) ICG fluorescence and tumour margins as defined at the microscopic level by the pathologist | 17 months

CONTACTS AND LOCATIONS:
Overall Officials: Danièle Noterman, MD, Principal Investigator — Jules Bordet Institute
Locations (1):
- Jules Bordet Institute, Brussels, Belgium